CLINICAL TRIAL: NCT05818488
Title: The Effect of a Mind-body Exercise Program on Aspects of Attention in Individuals With Anxiety: Protocol for a Randomized Controlled Trial
Brief Title: The Effect of a Mind-body Exercise Program on Aspects of Attention in Individuals With Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, Erica Simone Rodrigues Moraes, Master Student Mental Health, Universidade Federal do Rio de Janeiro
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IPUBBM
Record Dates: First submitted 2023-03-14; First posted 2023-04-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Anxiety Disorder
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental mind-body intervention (Experimental): subjects will be randomized into intervention (one session of mindbody exercise), where they will be asked to sit in a comfortable armchair and remain in a comfortable posture with eyes closed. Cognitive evaluation will be done before and after the intervention.
  Interventions: Other: Experimental mind-body intervention
- Control group (No Intervention): This group will be submitted to the same evaluation. However, they will wiat for 15 minutes with no intervention.

INTERVENTIONS:
Other: Experimental mind-body intervention — A meditation will be guided by an audio through headphones. The audio will last 15 minutes with an initial invitation to centering (full attention to the state of the body and the breath, bringing the attention to the present moment), followed by body scanning, followed by targeting the seven dimensions of interoceptive capacity (noticing, not being distracted, not worrying, attentional regulation, emotional awareness, self-regulation, and trust), and the passive control group (waiting room)
  Arms: Experimental mind-body intervention

SUMMARY:
Mind-body exercises is a non-pharmacological intervention to mental health and can improve interoceptive capacity. Interoceptive is linked to the process of sensory information within the body playing an important role in behavior. Consequently, interoceptive can be modulated by mind-body training through sustained attention to breathing signals, certainty of movements, and also related to activation of brain processes. The present study aimed to evaluation the effect of mind-body in interoceptive capacity in individuals with anxiety. An anamnesis will be performed with demographic data, as well as questions about medications and physical and mental health history. After that, subjects will be randomized into an intervention (one session of mind-body exercises) where they will be asked to sit in a comfortable armchair and remain in a comfortable posture with their eyes closed. A meditation will be guided by an audio through headphones. The audio will last 15 minutes with an initial invitation to centering (full attention to the state of the body and the breath, bringing the attention to the present moment), followed by a body scan considering the seven dimensions of interoceptive capacity (noticing, not being distracted, not worrying, attentional regulation, emotional awareness, self-regulation, and trust) and the passive control group (waiting room), after the intervention the same cognitive tests will be reapplied. Then, the groups will be switched for a crossover analysis.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of anxiety
* must be able to understand procedures

Exclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
interoceptive capacity. | 15 minutes after the intervention
  Evaluated by the interoceptive awareness multidimensional assessment scale, the average of each of the seven dimensions is calculated, the higher the value, the higher the interoceptive capacity
Anxiety symptoms | 15 minutes after the intervention
  A 14-item Hamilton anxiety scale will be applied, each item is scored from 0 (absent symptoms) to 4 (disabling symptoms)
Concentrated attention test | 15 minutes after the intervention
  The D2-R Concentrated Attention Assessment Test evaluates the ability to concentrate attention, realized by the speed and accuracy with which the individual can discriminate symbols.
  The test is composed of the letters d or p, and 1 to 4 strokes. In total, get 13 different signs, of which three (d with 2 dashes) represent the target objects, the task is to cancel all the target objects of the test (d with 2 dashes)
Digit Span test | 15 minutes after the intervention
  Assists in measuring the Distraction Resistance Index. The direct order is applied first applied first, followed by the reverse order, which is administered The direct order is applied first, followed by the reverse order, which is administered regardless if the examinee fails the direct order entirely.
  Each item is made up of two sets of digits constituting two trials, both of which are applied.
  attempts, both of which are applied. The maximum score on the subtest is 30 points, where the maximum raw score in direct order is 16 points while in reverse order it is 14 points.

IPD SHARING:
Plan to Share IPD: No